CLINICAL TRIAL: NCT03487393
Title: Determination of Threshold of Stimulation, Tolerability and Safety of Magnetic Nerve Stimulation In Healthy Subjects: an Exploratory Study
Brief Title: VitalFlow Healthy Volunteer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nervive, Inc. (Industry)
Collaborators: Centro Nacional de Investigacion en Imagenologia e Instrumentacion Medica (CI3M) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRV_PI_01_15
Record Dates: First submitted 2017-06-17; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Normal Subject / Healthy Volunteers
Keywords: facial nerve; magnetic stimulation; cerebral blood flow

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitalflow treatment (Experimental): The subject's exposure will be through a ramp model of increments in magnetic stimulation power delivered to the facial nerves bilaterally. Increases in magnetic stimulation will be 10% for 10 seconds from 10% to 60%. Subsequent to this will be evaluated for 5 minutes in the power of tolerability of the subject (60% 70%, 80% or 90%).
  Interventions: Device: magnetic facial nerve stimulation

INTERVENTIONS:
Device: magnetic facial nerve stimulation — Magnetic stimulation of facial nerve.

SUMMARY:
Find the stimulation threshold of the facial nerve (ganglion Geniculate) associated with tolerability and safety in subjects Healthy humans.

DETAILED DESCRIPTION:
Magnetic stimulation of the facial nerve (geniculate ganglion) in humans can induce changes in cerebral blood flow safely, without generating adverse effects unknown to the technique.

Our specific objectives:

1. Perform tolerability and safety tests of magnetic stimulation on the facial nerve.
2. Establish the optimal stimulation threshold associated with tolerability in order to apply it to the final design of the Magnetic Stimulation (MS) system.
3. Measure whether the threshold found shows any increase in cerebral perfusion in the subject with respect to their baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Normal audiometry chart (Evaluated at the time of your inclusion).
* Normal neurological examination at time of inclusion.

Exclusion Criteria:

* Subjects with a diagnosis of epilepsy, seizures, facial nerve palsy, migraine or recurrent headaches, glaucoma or neuropathies.
* Subjects in breastfeeding or in pregnancy. (To be confirmed with test strip).
* Subjects with acute or acute chronic medical conditions.
* Age less than 20 years or greater than 40 years.
* Carotid surgery.
* Episodes of syncope.
* Known arteriosclerosis anywhere on the body
* Metal implants (cochlear implants, pacemakers, metal prostheses).
* Intracranial abnormalities observed by MRI or MRA (Evaluated at time of inclusion of the subject).
* Intraocular pressure> 22mmHg (Evaluated at time of inclusion of the subject)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2016-01-08 (Actual)

PRIMARY OUTCOMES:
Change in perfusion index of cerebral blood flow | 10 minutes post-stimulation
  An algorithm to calculate the perfusion index using magnetic resonance images across the entire brain

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Nacional de Investigación en Imagenología e Instrumentación Medica, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
available from investigators authors upon reasonable request